CLINICAL TRIAL: NCT01551667
Title: Observational and Comparative Study on the Immune Response of Patients With Chronic, Staphylococcus Aureus-infected Wounds (Localized Infections Versus Bacteremia)
Brief Title: Immune Response of Patients With Chronic, Staphylococcus Aureus-infected Wounds
Acronym: ORISA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2011/JPL-02; 2011-A01400-41 (Other: RCB number)
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Diabetic Foot; Foot Ulcer; Leg Ulcer; Bacteremia; Infection
Keywords: S. aureus
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Leg Ulcer; Bacteremia; Infections; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Left over blood/serum/plasma specimens will be incorporated into the biobank at the Bacteriology Laboratory of the Nîmes University Hospital
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases / bacteraemia: Patients consulting at the departments of Diabetology, Dermatology or Infectious Diseases of the participating hospitals and who have (1) inaugural or recurrent diabetic foot/ankle ulcers of Grade 2-4, or (2) who have an infected leg ulcer (arterial, venous, or mixed. This infection must involve S. aureus in a mono-or polymicrobial setting. This group of patients has bacteraemia.
  Interventions: Biological: Antibody assays for S. aureus; Biological: Basic blood work
- Controls: Patients consulting at the departments of Diabetology, Dermatology or Infectious Diseases of the participating hospitals and who have (1) inaugural or recurrent diabetic foot/ankle ulcers of Grade 2-4, or (2) who have an infected leg ulcer (arterial, venous, or mixed. This infection must involve S. aureus in a mono-or polymicrobial setting. This group of patients does not have bacteraemia.
  Interventions: Biological: Antibody assays for S. aureus; Biological: Basic blood work

INTERVENTIONS:
Biological: Antibody assays for S. aureus — Antibody assays for S. aureus at Day 0, Day 2, Day 4, Day 7, Day 30 and Month 6.
Biological: Basic blood work — Hemogramme + CRP on Days 0, 2, 4 and 7

SUMMARY:
The primary objective of this study is to detect differences in anti-S. aureus antibody assays (IgM, IgA, IgG and its subclasses) between (1) a group of patients with bacteremia due to a chronic wound (cases) and (2) a group of patients with localized chronic wound infections (control).

DETAILED DESCRIPTION:
Secondary objectives include:

* To propose a diagnostic marker of bacteraemia based on the detection of anti-S. aureus by xMAP technology
* To evaluate the kinetics of the humoral immune response to S. aureus in patients with bacteraemia
* To evaluate the virulence of S. aureus isolated from chronic, infected wounds
* To enrich the Nîmes University Hospital biobank
* To evaluate the prevalence of different antibodies within each group

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 6 months of follow up
* Patients consulting at the departments of Diabetology, Dermatology or Infectious Diseases of the participating hospitals
* inaugural or recurrent diabetic foot/ankle ulcers of Grade 2-4, or (2) who have an infected leg ulcer (arterial, venous, or mixed.

Controls:

* Absence of bacteriemia

Cases:

* Presence of bacteriemia

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient does not have a chronic wound
* Patient with grand 1 ulcer
* Patient's wound/ulcer is not infected
* Patient's would/ulcer is infected, but not involving S. aureus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting at the departments of Diabetology, Dermatology or Infectious Diseases of the participating hospitals and who have (1) inaugural or recurrent diabetic foot/ankle ulcers of Grade 2-4, or (2) who have an infected leg ulcer (arterial, venous, or mixed). This infection must involve S. aureus in a mono-or polymicrobial setting.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2012-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Humoral immune response | 6 months
  Humoral immune response via production of anti-staphylococci antibodies in patients with bacteraemia versus those with localized wound infections. 22 antibodies will be tested(quantitative determination by xMAP technology).

SECONDARY OUTCOMES:
Antibody production kinetics | 6 months
  Kinetics of the production of the 22 antibodies against S. aureus in the 2 groups. The temporal evolution of antibody titres determined via xMAP technology will be followed throughout the study.
Presence / absence of clonal complexes of the S. aureus strains | 6 months
  determined by microarrays

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Lavigne, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (6):
- France (6):
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard
  - CHU de Nîmes - Hôpital Universitaire de Réadaptation du Grau du Roi, Le Grau-du-Roi
  - CHU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - CHU de Nantes - Hôtel-Dieu, Nantes
  - CHU de Nice - Hôpital Pasteur, Nice
  - CHU de Nice - Hôpitaux L'Archet 1 et 2, Nice